CLINICAL TRIAL: NCT05351567
Title: The Effect of The Educatıonal Program Created Accordıng to Transformatıonal Learnıng Theory on Infertılıty and Stigma in Infertılıty Women
Brief Title: Transformatıonal Learnıng Theory on Infertılıty and Stigma in Infertılıty Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Şengül Yaman Sözbir, Prof. dr., Gazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 77082166-604
Record Dates: First submitted 2022-03-31; First posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Infertility, Female; Stigma, Social
Keywords: infertility; stigma; educatiıon
MeSH Terms: conditions — Infertility, Female; Social Stigma; Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- infertility educatıon group (Experimental): women wıll educate with model about infertility
  Interventions: Other: EDUCATIONAL PROGRAM CREATED ACCORDING TO TRANSFORMATIONAL LEARNING THEORY
- control group (non-education) (No Intervention): Routıne care

INTERVENTIONS:
Other: EDUCATIONAL PROGRAM CREATED ACCORDING TO TRANSFORMATIONAL LEARNING THEORY — EDUCATIONAL PROGRAM CREATED ACCORDING TO TRANSFORMATIONAL LEARNING THEORY FOR INFERTILITY FEMALES
  Arms: infertility educatıon group

SUMMARY:
This study will be conducted to evaluate the effect of the education program created according to the transformational learning theory on women being affected by infertility and feeling stigmatized due to infertility.

The research is a single center parallel group simple randomized controlled trial. The sample consisted of 52 participants in total.

determined to be formed. Diagnosed with infertility, literate, 18 years of age and older, no communication disability, and Women who volunteer to participate will be included in the study. Personal Information Form, Infertility Affected Scale and Infertility Stigma (Stigma) Scale will be used to collect data. Groups of 3-10 people were formed for the women in the experimental group.

A training program consisting of four modules will be implemented once a week. Data analysis in SPSS 22.0 package program will be.

DETAILED DESCRIPTION:
Nurses have important duties in providing counseling and support to infertile individuals during this crisis, which is very difficult to cope with. In this context, nurses should provide psychosocial care that will enable the individual to accept and cope with the current process. This study will be conducted to evaluate the effect of the education program created according to the transformational learning theory on women being affected by infertility and feeling stigmatized due to infertility. The study was planned as a single-center parallel group simple randomized controlled trial. The population of the study will be women who applied to Tatvan Maternity and Children's Hospital due to infertility between 22/05/2022-22/05/2023. Power analysis was performed to determine the number of samples. For this, the information in a similar study (Infertility Stigma Scale Experiment Mean: 38.67±4.75, Control Mean: 69.76±4.5) was used as a reference. Analysis was done in G power version 3.1. The minimum number of participants required to be included in each group was determined as 22, with a total of 44 (α=0.05, 1-β=0.95). However, considering the loss rate (21.77%) in the reference study, the total number of participants was increased by 20% to 52 (experimental: 26, control: 26). Personal Information Form, Infertility Affected Scale and Infertility Stigma (Stigma) Scale will be used to collect data. Application First of all, the aim and content of the research will be explained to the women. Their compliance with the sampling inclusion criteria will be evaluated. Afterwards, women who agreed to participate in the study will have an informed consent form signed. Personal information form and pre-tests (Infertility Affect Scale and Infertility Stigma Scale) will be applied to women. Then, the women will be randomly randomized to assign the experimental and control groups. Contact information (Phone numbers and e-mail addresses) will be taken at the first encounter.

Experimental Group Application

A training program consisting of four modules created according to Transformational Learning Theory will be applied once a week to the women in the experimental group by forming groups of 3-10 people. Post-tests (Infertility Affect Scale and Infertility Stigma Scale) will be applied within 1 week after the training is over and in the 4th week after that. The training modules and the training methods to be used in the modules are given below:

Module 1: Infertility Based on Gender Patterns: Meaning structures of "femininity", "motherhood" and "infertility" in society Dating activity, brainstorming, discussion over experiences, critical reflection Module 2: Violence due to infertility (The Concept of Stigma): Domestic and Social Pressure/Violence Introductory activity, role-play, sharing feelings, discussion over experiences, critical reflection Module 3: Punishment and exposure to traditional practices for infertility Introductory activity, watching the movie, interpreting the movie through experiences, critical reflection Module 4: Interpreting the awareness experienced in the education process and sharing future plans Introductory activity, presentation (by women), peer review Control group application The post-tests (Infertility Affect Scale and Infertility Stigma Scale) will be applied to the women in the control group 5 weeks after the pre-test application and 4 weeks after this application.

ELIGIBILITY:
Inclusion criteria for research;

* Being diagnosed with infertility
* Being at least literate
* Be at least 18 years old
* Not having a communication barrier
* Volunteering to participate in the research Exclusion Criteria from the Sample;
* The woman's desire to withdraw from the research
* Not filling out data collection tools
* Unable to reach for training/consulting

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-05-15 (Estimated); Primary Completion 2023-05-15 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
change between the mean score of the Infertility Affected Scale of infertile women who participated in the training program created according to the transformative learning theory and who did not. | 9 weeks
  Infertility Affect Scale
change between the mean score of the Infertility Stigma (Stigma) Scale of infertile women who participated and did not participate in the training program created according to the transformative learning theory. | 9 weeks
  Infertility Stigma (Stigma) Scale

CONTACTS AND LOCATIONS:
Overall Officials: Sıdıka PELİT AKSU, PhD, Principal Investigator — Gazi University

IPD SHARING:
Plan to Share IPD: No